CLINICAL TRIAL: NCT02738541
Title: Evaluation of Anti-calculus Efficacy of a Dentrifice Containing Sodium Pyrophosphate and Potassium Pyrophosphate in Heavy Calculus Formers
Brief Title: Anti-calculus Efficacy of a Dentrifice Containing Sodium Pyrophosphate and Potassium Pyrophosphate in Heavy Calculus Formers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Government Dental College and Research Institute, Bangalore (Other)
Responsible Party: Principal Investigator, Dr. A R Pradeep, Professor & Head, Department of Periodontology, Government Dental College and Research Institute, Bangalore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GDCRI/ACM/PG/PhD/2/2014-2015FN
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: ANTICALCULUS EFFICACY OF PYROPHOSPHATE IN HEAVY CALCULUS FORMERS
MeSH Terms: interventions — Sodium

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Group 1 (Active Comparator): DENTRIFICE CONTAINING 5% SODIUM AND POTASSIUM PYROPHOSPHATE WAS PRESCRIBED AND SUBJECTS WERE EVALUATED AT 3MONTH AND 6 MONTHS
  Interventions: Drug: DENTRIFICE CONTAINING 5% SODIUM AND POTASSIUM PYROPHOSPHATE
- Group 2 (Placebo Comparator): PLACEBO DENTRIFICE WITHOUT PYROPHOSPATE WAS PRESCRIBED AND SUBJECTS WERE EVALUATED AT 3MONTH AND 6 MONTHS
  Interventions: Drug: PLACEBO DENTRIFICE WITHOUT PROPHOSPHATE

INTERVENTIONS:
Drug: DENTRIFICE CONTAINING 5% SODIUM AND POTASSIUM PYROPHOSPHATE — DENTRIFICE CONTAINING 5% SODIUM AND POTASSIUM PYROPHOSPHATE WAS ADVISED TWICE DAILY FOR 6 MONTHS
  Other Names: XTAR
  Arms: Group 1
Drug: PLACEBO DENTRIFICE WITHOUT PROPHOSPHATE — PLACEBO DENTRIFICE WITHOUT PYROPHOSPHATE WAS ADVISED TWICE DAILY FOR 6 MONTHS
  Arms: Group 2

SUMMARY:
The purpose of this study was to determine the anti-calculus effect of dentrifice containing 5% sodium pyrophosphate and potassium pyrophosphate in a triple-mask placebo controlled randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 15-30 years.
2. Subjects who have not received periodontal therapy within preceding 1year.
3. Heavy calculus formers with simplified calculus index score 1.5-3 .

Exclusion Criteria:

1. Age group 15-30 years.
2. Subjects who have not received periodontal therapy within preceding 1year.
3. Heavy calculus formers with simplified calculus index score 1.5-3 .

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
simplied calulus index. | Baseline to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Government Dental College and Research Institute, Bangalore, Karnataka, India